CLINICAL TRIAL: NCT04758416
Title: A Phase II, Single-center STudy on the vAlue of Non-invasive Dual-Pet（18F-FES PET and 68Ga-HER2-Affibody PET）InformatiOn IN Subtype of Metastatic Breast Cancer(MBC)
Brief Title: Study on the Value of Non-invasive Dual-Pet Information in Subtype of Metastatic Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Director of department of medical oncology, Fudan University
Other Study IDs: STANDPOINT
Record Dates: First submitted 2021-02-14; First posted 2021-02-17 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy; 16-fluoroestradiol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic breast cancer patients: 50 metastatic breast cancer patients
  Interventions: Procedure: biopsy or surgical pathology in metastases; Drug: 68Ga-HER2 affibody,18F-FDG, 18F-FES

INTERVENTIONS:
Procedure: biopsy or surgical pathology in metastases — biopsy or surgical pathology in extrahepatic/liver/brain metastases
Drug: 68Ga-HER2 affibody,18F-FDG, 18F-FES — 68Ga-NOTA-MAL-MZHER2 (68Ga-HER2) affibody is an investigational Positron Emission Tomography (PET)/ Computed Tomography (CT) radiopharmaceutical.

SUMMARY:
Study on the Value of Non-invasive Dual-Pet(18F-FES PET and 68Ga-HER2-Affibody PET) Information in Subtype of Metastatic Breast Cancer

DETAILED DESCRIPTION:
A Phase II, Single-center STudy on the vAlue of Non-invasive Dual-Pet（18F-FES PET and 68Ga-HER2-Affibody PET）InformatiOn IN Subtype of Metastatic Breast Cancer(MBC)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily joined the study, signed informed consent, and had good compliance.
2. Female patients aged over 18 years (including cutoff value).
3. an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
4. Recurrence or metastatic breast cancer confirmed by histopathology, or expect to be feasible metastasis puncture or surgery to confirm histopathological recurrence or metastatic breast cancer.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Alcohol allergy is not suitable for FES-PET/ C.
3. There are contraindications for patients who are expected to have metastasis puncture or surgery.
4. Mental disorders or other conditions affecting patient compliance.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 metastatic breast cancer patients
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Verify the subtype value of dual-PET in extrahepatic metastases | 2 year
  Verify whether the subtype value of FES-PET and HER2-PET is consistent with biopsy or surgical pathology in extrahepatic metastases.

SECONDARY OUTCOMES:
Verify the HER2-PET value in liver metastasis | 2 year
  Verify whether the HER2-PET value is consistent with biopsy or surgical pathology in liver metastasis.
Verify the HER2-PET value in brain metastasis | 2 year
  Verify whether the HER2-PET value is consistent with biopsy or surgical pathology in brian metastasis.
Heterogeneity in metastatic lesions | 2 year
  Observe the heterogeneity of ER and HER2 expression in metastatic lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Shanghai Cancer Center Institutional Review Board, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No